CLINICAL TRIAL: NCT05184231
Title: Patient and Physician Survey on Satisfaction With Somatostatin Analogue (SSA) Injections in Acromegaly in China
Status: Withdrawn | Type: Observational
Why Stopped: Study wasn't feasible anymore. It was withdrawn on 13 Jan 2023.
Sponsor: Ipsen (Industry)
Responsible Party: Sponsor
Other Study IDs: CLIN-52030-454
Record Dates: First submitted 2021-12-23; First posted 2022-01-11 (Actual); Last update posted 2023-03-17 (Actual); Status verified 2023-03

CONDITIONS: Acromegaly
MeSH Terms: conditions — Acromegaly

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Patient cohort
- Physician cohort

SUMMARY:
The purpose of the protocol is to achieve an in-depth understanding of the current satisfaction status of somatostatin analogue (SSA) treatment for acromegaly through patient and physician surveys.

ELIGIBILITY:
Inclusion Criteria:

For Patients:

* Age 18 years or older
* Diagnosed with acromegaly
* Receiving current SSA injections for acromegaly treatment for at least 3 months
* Signed electronic Informed Consent Form (eICF)

For Physicians:

* Licensed endocrinologists or neurosurgeons
* Having prescribed SSAs for at least five patients with acromegaly in the past 6 months
* Signed eICF

Exclusion Criteria:

* Patients will not be included in the survey if they meet any of the following criteria:
* Patients who are not able to successfully complete the questionnaire independently
* Pregnant patients

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Primary care clinic
Sampling Method: Non-Probability Sample
Enrollment: 0 (Actual)
Dates: Start 2023-02-13 (Estimated); Primary Completion 2023-10 (Estimated); Study Completion 2023-10 (Estimated)

PRIMARY OUTCOMES:
Overall patient satisfaction with SSA treatment. | During the whole study period (approximately 3 months).
  To be assessed by four levels of satisfaction including very satisfied, satisfied, dissatisfied, and very dissatisfied

SECONDARY OUTCOMES:
Patient satisfaction with symptom control of SSA treatment | During the whole study period (approximately 3 months).
Patient satisfaction with frequency of administration of SSA treatment | During the whole study period (approximately 3 months).
Patient satisfaction with mode of administration of SSA treatment | During the whole study period (approximately 3 months).
Patient satisfaction with convenience of administration of SSA treatment | During the whole study period (approximately 3 months).
Patient satisfaction with injection site reactions of SSA treatment | During the whole study period (approximately 3 months).
Patient satisfaction with adverse reactions to SSA treatment | During the whole study period (approximately 3 months).
Physician overall satisfaction with SSA treatment. | During the whole study period (approximately 3 months).
  The satisfaction rate is calculated as the proportion of physicians who reported to be satisfied or very satisfied with the prescribed SSA treatment.
Physician satisfaction with symptom control of SSA treatment | During the whole study period (approximately 3 months).
Physician satisfaction with frequency of administration of SSA treatment | During the whole study period (approximately 3 months).
Physician satisfaction with mode of administration of SSA treatment | During the whole study period (approximately 3 months).
Physician satisfaction with convenience of administration of SSA treatment | During the whole study period (approximately 3 months).
Physician satisfaction with injection site reactions of SSA treatment | During the whole study period (approximately 3 months).
Physician satisfaction with adverse reactions to SSA treatment | During the whole study period (approximately 3 months).
Aspects of patient concern before initiating SSA treatment | During the whole study period (approximately 3 months).
  The magnitude of concern will be assessed by four levels including not concerned, slightly concerned, concerned, and very concerned.
Aspects of physician concern before prescribing SSA treatment | During the whole study period (approximately 3 months).
  The magnitude of concern will be assessed by four levels including not concerned, slightly concerned, concerned, and very concerned.
Overall patient satisfaction with SSA treatment: satisfied versus dissatisfied with their SSA treatment. | During the whole study period (approximately 3 months).
  The patient satisfaction will be categorized as binary variables including satisfied (very satisfied and satisfied) versus dissatisfied (dissatisfied and very dissatisfied).

IPD SHARING:
Plan to Share IPD: Yes
Qualified researchers may request access to patient level data and related study documents including the clinical study report, study protocol with any amendments, annotated case report form, statistical analysis plan, and dataset specifications. Patient level data will be anonymized and study documents will be redacted to protect the privacy of study participants.
  Any requests should be submitted to www.vivli.org for assessment by an independent scientific review board.
Time Frame: Where applicable, data from eligible studies are available 6 months after the studied medicine and indication have been approved in the US and EU or after the primary manuscript describing the results has been accepted for publication, whichever is later.
Access Criteria: Further details on Ipsen's sharing criteria, eligible studies and process for sharing are available here (https://vivli.org/members/ourmembers/)
URL: https://vivli.org/members/ourmembers/